CLINICAL TRIAL: NCT02244645
Title: Effects of Yoga Versus Passive Modality on Pain, Disability, Salivary Cortisol Concentrations, Brain- Derived Neurotropic Factor, Heart Rate Variability and Immune Functions Among Patients With Chronic Low Back Pain: A Randomized Controlled Trial
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Chang Bing Show Chwan Memorial Hospital (Other)
Responsible Party: Principal Investigator, Shu-Hui Yeh, RN, PhD, Professor, Chang Bing Show Chwan Memorial Hospital
Allocation: Randomized | Model: Parallel | Masking: Single
Other Study IDs: 1010803
Record Dates: First submitted 2014-09-16; First posted 2014-09-19 (Estimated); Last update posted 2014-09-19 (Estimated); Status verified 2014-09

CONDITIONS: Low Back Pain
Keywords: Low back pain, physical therapy, yoga.
MeSH Terms: conditions — Low Back Pain

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Passive modality control group (Other): Passive modality control group will receive regular 40-minutes rehabilitation twice a week for 3 months.
  Interventions: Behavioral: passive modality
- Yoga treatment group (Experimental): Yoga treatment group will receive regular 60-minutes yoga classes twice a week for 4 months.
  Interventions: Behavioral: Yoga treatment

INTERVENTIONS:
Behavioral: passive modality — Passive modality control group will receive regular 40-minutes rehabilitation twice a week for 3 months.
  Arms: Passive modality control group
Behavioral: Yoga treatment — Yoga treatment group will receive regular 60-minutes yoga classes twice a week for 4 months.
  Arms: Yoga treatment group

SUMMARY:
This study may clarify a potential promising mechanism and clearest evidence to support the value of yoga as a therapeutic option for reducing chronic low back pain.

DETAILED DESCRIPTION:
Low back pain is a common problem, with 70-80% of adults were bothered in their lives, which influence the work and quality of life. Yoga is one of the most popular complementary and alternative medicine for back pain, and this mind-body intervention has increasingly chosen to effectively treat chronic pain.

This is a parallel-arm randomized controlled trial which will compare the outcomes of participants assigned to the experimental treatment group (yoga, with 36 participants) with those assigned to a passive modality control group for 3 months (12 weeks). Each group will receive regular 60-minutes yoga classes or passive modality twice a week. The investigators confer the difference of pain relief and functional life improvement between passive modality and yoga. The latter is expected to have positive effects on Chronic low back pain. The effects and possible mechanisms of action responsible for passive modality and yoga on salivary cortisol concentrations, inflammatory cytokines and autonomic nervous tone will be also evaluated. The study's primary endpoints are (1) back pain relief, (2) functional life improved, (3) Salivary cortisol concentrations decreased, (4) brain-derived neurotrophic factor improved, (5) heart rate variability improved, and (6) immune function improved significantly among the participants in the experimental group than the control group.

This study may clarify a potential promising mechanism and clearest evidence to support the value of yoga as a therapeutic option for reducing chronic low back pain. If the results are positive, clinicians will attain more options for treating patient with chronic low back. Furthermore, the positive results from this study will help focus more future in-depth research on the most promising potential mechanism of action identifies.

ELIGIBILITY:
Inclusion Criteria:

* Patient with idiopathic low back pain of more than 12 weeks.

Exclusion Criteria:

* Current pregnancy
* Diagnosis of ankylosing spondylitis, osteoporosis, fibromyalgia, failed back syndrome and other chronic illnesses.
* Inability to participate yoga exercise regularly.
* Accept steroid treatment within 3 months.
* BMI > 30

Ages: 20 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 86 (Estimated)
Dates: Start 2013-12; Primary Completion 2015-11 (Estimated); Study Completion 2015-11 (Estimated)

PRIMARY OUTCOMES:
Back pain relief and functional life improved | Change from baseline in back pain and life quality at 6 months
  Back pain relief and functional life improved will assessed by visual analogue scale (VAS) and Roland-Morris disability questionnaire at five different times: (1)baseline data : before intervention, (2)outcome data: 3, 6, 9 and 12 week yoga exercise, right after exercise measure post-test.

SECONDARY OUTCOMES:
Salivary cortisol concentrations decreased | Change from baseline in salivary cortisol at 6 months
  Cortisol concentrations will be measured at three different times: (1)baseline data : before intervention, (2)outcome data: 6 and 12 week yoga exercise, right after exercise measure post-test.
Heart rate variability improved | Change from baseline in heart rate variability at 6 months
  Heart rate variability will be measured at three different times: (1)baseline data : before intervention, (2)outcome data: 6 and 12 week yoga exercise, right after exercise measure post-test.
Immune function improved | Change from baseline in immune function at 6 months
  Immune function will be assessed by blood analysis including lymphocyte subpopulations (Th1/ Th2/ Treg/ Th17), polarization (T-bet/ Gata-3/ Foxp3/ RORrt), its related cytokines (Th1: IL-12/ IFN-γ/ IL-27; Th2: IL-4/ IL-13/ IL-25; Th17: IL-17A/ IL-6/ IL-21; Treg: TGF/ IL-10), lipid prolife and C-reactive protein at at three different times: (1)baseline data : before intervention, (2)outcome data: 6 and 12 week yoga exercise, right after exercise measure post-test.
Brain-derived neurotrophic factor improved | Change from baseline in brain-derived neurotrophic factor at 6 months
  Brain-derived neurotrophic factor will be assessed by blood analysis at at three different times: (1)baseline data : before intervention, (2)outcome data: 6 and 12 week yoga exercise, right after exercise measure post-test.

CONTACTS AND LOCATIONS:
Overall Officials: Kuender D. Yang, MD, PhD, Study Chair — Chang Bing Show Chwan Memorial Hospital; Shu-Hui Yeh, PhD., Study Director — Chang Bing Show Chwan Memorial Hospital; Kwan-Yu Chan, MD., Principal Investigator — Chang Bing Show Chwan Memorial Hospital
Locations (1):
- Division of Core Laboratory; Chang Bing Show Chwan Memorial Hospital, Changhua County, Taiwan